CLINICAL TRIAL: NCT03468426
Title: An Open Label Phase Ib Dose Finding Study of BI 836880 in Combination With Ezabenlimab to Characterize Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy in Patients With Locally Advanced or Metastatic Non-squamous Non-Small Cell Lung Cancer and in Other Solid Tumors
Brief Title: A Study to Test Different Doses of BI 836880 Combined With Ezabenlimab in Patients With Advanced Non-small Cell Lung Cancer Followed by Other Types of Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1336-0011; 2017-001378-41 (EudraCT Number)
Record Dates: First submitted 2018-03-08; First posted 2018-03-16 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Non-squamous, Non-Small-Cell Lung Cancer; Neoplasms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Part 1 - BI 836880 360 mg (Experimental): Patients with locally advanced or metastatic non-squamous non-small cell lung cancer (NSCLC) who progressed during or after first line platinum-based chemotherapy, received 360 milligram (mg) BI 836880 and 240 mg Ezabenlimab (BI 754091) as an intravenous infusion on day 1 of each 3-week cycle until progression, unacceptable toxicity, or up to a maximum of 53 cycles.
  Interventions: Drug: BI 836880; Drug: Ezabenlimab
- Part 1 - BI 836880 500 mg (Experimental): Patients with locally advanced or metastatic non-squamous non-small cell lung cancer (NSCLC) who progressed during or after first line platinum-based chemotherapy, received 500 milligram (mg) BI 836880 and 240 mg Ezabenlimab (BI 754091) as an intravenous infusion on day 1 of each 3-week cycle until progression, unacceptable toxicity, or up to a maximum of 53 cycles.
  Interventions: Drug: BI 836880; Drug: Ezabenlimab
- Part 1 - BI 836880 720 mg (Experimental): Patients with locally advanced or metastatic non-squamous non-small cell lung cancer (NSCLC) who progressed during or after first line platinum-based chemotherapy, received 720 milligram (mg) BI 836880 and 240 mg Ezabenlimab (BI 754091) as an intravenous infusion on day 1 of each 3-week cycle until progression, unacceptable toxicity, or up to a maximum of 53 cycles.
  Interventions: Drug: BI 836880; Drug: Ezabenlimab
- Part 2 - Cohort A, 2nd line NSCLC (Experimental): Patient with pathologically confirmed locally advanced or metastatic non-squamous NSCLC who progressed during or after check-point inhibitor monotherapy treatment. Patient must also have received treatment with a platinum-based chemotherapy regimen and have progressed or be intolerant, or ineligible, as per applicable local practice. Patients received 720 milligram (mg) BI 836880 and 240 mg Ezabenlimab (BI 754091) as an intravenous infusion on day 1 of each 3-week cycle until progression, unacceptable toxicity, or up to a maximum of 53 cycles.
  Interventions: Drug: BI 836880; Drug: Ezabenlimab
- Part 2 - Cohort B, 3rd line NSCLC (Experimental): Patient with pathologically confirmed locally advanced or metastatic non-squamous NSCLC who progressed during or after platinum-based chemotherapy and a check-point inhibitor (CPI) combination treatment as the most recent anticancer treatment. Patients received 720 milligram (mg) BI 836880 and 240 mg Ezabenlimab (BI 754091) as an intravenous infusion on day 1 of each 3-week cycle until progression, unacceptable toxicity, or up to a maximum of 53 cycles.
  Interventions: Drug: BI 836880; Drug: Ezabenlimab
- Part 2 - Cohort C, SCLC (Experimental): Patient with pathologically confirmed locally advanced or metastatic Small Cell Lung Cancer (SCLC) with documented intolerance to platinum-based chemotherapy or refractory to platinum-based chemotherapy. Patients who were platinumsensitive must also have received one additional prior line of platinum-based chemotherapy, if eligible, with or without combination with CPI as per applicable local treatment country guidelines. Patients received 720 milligram (mg) BI 836880 and 240 mg Ezabenlimab (BI 754091) as an intravenous infusion on day 1 of each 3-week cycle until progression, unacceptable toxicity, or up to a maximum of 53 cycles.
  Interventions: Drug: BI 836880; Drug: Ezabenlimab
- Part 2 - Cohort D, glioblastoma (Experimental): Patient with histologically confirmed recurrent glioblastoma with no more than two previous lines of chemotherapy. Patients received 720 milligram (mg) BI 836880 and 240 mg Ezabenlimab (BI 754091) as an intravenous infusion on day 1 of each 3-week cycle until progression, unacceptable toxicity, or up to a maximum of 53 cycles.
  Interventions: Drug: BI 836880; Drug: Ezabenlimab
- Part 2 - Cohort E, Melanoma (Experimental): Patient with histologically confirmed, unresectable, Stage IV metastatic melanoma who progressed during or after CPI based regimen. Patients with a BRAF mutation must have received targeted treatment, or were not eligible, with a BRAF and MEK inhibitor as per applicable local country guidelines. Patients received 720 milligram (mg) BI 836880 and 240 mg Ezabenlimab (BI 754091) as an intravenous infusion on day 1 of each 3-week cycle until progression, unacceptable toxicity, or up to a maximum of 53 cycles.
  Interventions: Drug: BI 836880; Drug: Ezabenlimab
- Part 2 - Cohort F, 2nd line Hepatocellular Carcinoma (Experimental): Patient with locally advanced or metastatic and/or unresectable Hepatocellular Carcinoma (HCC) who were intolerant or progressed during 1st line sorafenib or lenvatinib treatment. Patients received 720 milligram (mg) BI 836880 and 240 mg Ezabenlimab (BI 754091) as an intravenous infusion on day 1 of each 3-week cycle until progression, unacceptable toxicity, or up to a maximum of 53 cycles.
  Interventions: Drug: BI 836880; Drug: Ezabenlimab
- Part 2 - Cohort G, 1st line Hepatocellular Carcinoma (HCC) (Experimental): Patient with locally advanced or metastatic and/or unresectable HCC with no prior systemic treatment. This will be implemented only in countries where this cohort is approved. Patients received 720 milligram (mg) BI 836880 and 240 mg Ezabenlimab (BI 754091) as an intravenous infusion on day 1 of each 3-week cycle until progression, unacceptable toxicity, or up to a maximum of 53 cycles.
  Interventions: Drug: BI 836880; Drug: Ezabenlimab
- Part 2 - Cohort H, 2nd line HCC - atezolizumab in combination with bevacizumab failures (Experimental): Patient with locally advanced or metastatic and/or unresectable Hepatocellular Carcinoma (HCC) who were intolerant or progressed during 1st line treatment with atezolizumab in combination with bevacizumab. Patients received 720 milligram (mg) BI 836880 and 240 mg Ezabenlimab (BI 754091) as an intravenous infusion on day 1 of each 3-week cycle until progression, unacceptable toxicity, or up to a maximum of 53 cycles.
  Interventions: Drug: BI 836880; Drug: Ezabenlimab

INTERVENTIONS:
Drug: BI 836880 — BI 836880 as an intravenous infusion on day 1 of each 3-week cycle.
Drug: Ezabenlimab — 240 mg Ezabenlimab (BI 754091) as an intravenous infusion on day 1 of each 3-week cycle.
  Other Names: BI 754091

SUMMARY:
This study has 2 parts. The first part was open to adults with advanced non-small cell lung cancer. The second part was open also to adults with other types of advanced cancer of the lung, brain, skin, and liver. After early encouraging results, more people with liver cancer can now take part in the study. The participants get a combination of two medicines called BI 836880 and ezabenlimab.

BI 836880 is a type of an antibody that blocks new blood vessel formation. New blood vessels are needed by the tumour to continue growing. Ezabenlimab is an antibody that may help the immune system fight cancer (immune checkpoint inhibitor).

The purpose of the first part of the study was to find out the highest dose of the BI 836880 that the participants can tolerate in combination with BI 754091. After the best dose of BI 836880 for the combination with ezabenlimab was found, it is used in the second part of the study. The purpose of the second part is to see whether the combination of BI 836880 and BI 754091 is able to make tumours shrink.

The participants are in the study as long as they benefit from and can tolerate treatment. During this time, they get infusions of BI 836880 and ezabenlimab every 3 weeks. The doctors also regularly check the general health of the participants.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* Of full age (according to local legislation, usually ≥ 18 years) at screening.
* Pathologically confirmed locally advanced or metastatic non-squamous NSCLC with PDL-1 expression available and >1% by IHC (as defined by the Pembrolizumab companion diagnostic test, determined by appropriate local pathology lab.
* No previous treatment with check-point inhibitor. Or patients with checkpoint inhibitor based treatment as last therapy before entering the trial.
* Documented disease progression or relapse (based on investigator's assessment) during or after completion of at least 2 cycles of platinum-based chemotherapy as first line treatment of Stage IIIB/IV non- squamous NSCLC or for checkpoint inhibitor experienced patients during or after completion of at least 2 cycles of platinum-based chemotherapy and a checkpoint inhibitor treatment (monotherapy or in combination with chemotherapy). This includes patients relapsing within 6 months of completing (neo)adjuvant/curative-intent chemotherapy/CPI or chemoradiotherapy
* At least one target lesion (outside the brain) that can be accurately measured per Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1 .
* Lesion with a diameter ≥ 2cm assessed by radiologist as suitable for DCE-MRI evaluation (Mandatory in Part 1, optional in Part 2)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 Life expectancy ≥ 3 months after start of the treatment in the opinion of the investigator
* Recovery from all reversible adverse events of previous anti-cancer therapies to baseline or CTCAE grade 1, except for alopecia (any grade), sensory peripheral neuropathy , must be ≤ CTCAE grade 2 or considered not clinically significant.
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
* Availability and willingness to provide a fresh tumour tissue sample obtained at baseline, and after 2 cycles of treatment
* Adequate organ function defined as all of the following (all screening labs should be performed at local lab within 10 days prior to treatment initiation)
* Male or female patients. Women of childbearing potential (WOCBP)1 and men able to father a child must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly, starting with the screening visit and through 6 months after the last dose of BI 836880 and BI 754091 treatment, respectively. A list of contraception methods meeting these criteria is provided in the patient information Note: Female patients of childbearing potential must have a negative serum pregnancy test within 72 hours prior to taking study medication during the screening period. At the following visits according to the flowchart a urine and/or serum pregnancy test is required. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. The serum pregnancy test must be negative for the patient to be eligible.

Part 2:

* Of full age (according to local legislation, usually ≥ 18 years) at screening
* At least one measurable target lesion outside the brain (excluding the glioblastoma patients where brain lesions are allowed), that can be accurately measured per RECIST version 1.1 or Response Assessment in Neuro-Oncology (RANO)
* ECOG performance status ≤ 1 (For glioblastoma cohort Karnofsky status is applicable)
* Adequate organ function as all of the following (all screening labs should be performed at local lab within approximately 72 hours prior to treatment initiation)
* Availability and willingness to provide a fresh tumor tissue sample obtained after relapse or progression on or after prior therapy. For Part 2, In case a fresh biopsy cannot be obtained (e.g. inaccessible lesions or patient safety concern), an archived specimen obtained up to 6 months prior to cycle 1, visit 1 (C1V1) may be submitted in case no systemic antineoplastic therapy has been administered between the biopsy and C1V1 (except for cohort D). For cohorts E, F and G, a fresh on-treatment biopsy is mandatory at C3D1, if possible from the same lesion as the pre-treatment biopsy.
* Life expectancy ≥ 3 months after start of the treatment in the opinion of the investigator
* Recovery from all reversible adverse events of previous anti-cancer therapies to baseline or CTCAE grade 1, except for alopecia (any grade), sensory peripheral neuropathy , must be ≤ CTCAE grade 2 or considered not clinically significant.
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
* Male or female patients. Women of childbearing potential (WOCBP)2 and men able to father a child must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly, for the entire duration of the trial treatment intake and for 6 months after the end of the trial treatment. A list of contraception methods meeting these criteria is provided in the patient information.

Note: Female patients of childbearing potential must have a negative serum pregnancy test within 72 hours during the screening period. At the following visits according to the flowchart, a urine and/or serum pregnancy test is required. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. The serum pregnancy test must be negative for the patient to be eligible.- Further inclusion criteria apply

Exclusion criteria:

Part 1:

* Known hypersensitivity to the trial drugs or their excipients or risk of allergic of anaphylactic reaction to drug product according to Investigator judgement (e.g. patient with history of anaphylactic reaction or autoimmune disease that is not controlled by nonsteroidal anti-inflammatory drugs (NSAIDs), inhaled corticosteroids, or the equivalent of </= 10 mg/day prednisone).
* Known immunodeficiency virus infection or an active hepatitis B or C virus infection.
* History of severe hypersensitivity reactions to other mAbs.
* Immunosuppressive corticosteroid doses (> 10 mg prednisone daily or equivalent) within 4 weeks prior to the first dose of trial medication.
* Current or prior treatment with any systemic anti-cancer therapy either within 28 days or a minimum of 5 half-lives, whichever is shorter before start of treatment.
* Serious concomitant disease, especially those affecting compliance with trial requirements or which are considered relevant for the evaluation of the endpoints of the trial drug, such as neurologic, psychiatric, infectious disease or active ulcers (gastrointestinal tract, skin) or laboratory abnormality that may increase the risk associated with trial participation or trial drug administration, and in the judgment of the investigator would make the patient inappropriate for entry into the trial.
* Major injuries and/or surgery or bone fracture within 4 weeks of start of treatment, or planned surgical procedures during the trial period.
* Patients with personal or family history of QT prolongation and/or long QT syndrome, or prolonged QTcF at baseline (> 480 ms).
* Significant cardiovascular/cerebrovascular diseases (i.e. uncontrolled hypertension, unstable angina, history of infarction within past 6 months, congestive heart failure > NYHA II).

Uncontrolled hypertension defined as: Blood pressure in rested and relaxed condition >= 140 mmHg, systolic or >= 90 mmHg diastolic (with or without medication), measured according to Appendix 10.2.

* LVEF < 50%
* History of severe hemorrhagic or thromboembolic event in the past 12 months (excluding central venous catheter thrombosis and peripheral deep vein thrombosis).
* Known inherited predisposition to bleeding or to thrombosis in the opinion of the investigator.
* Patient with brain metastases that are symptomatic and/or require therapy.
* Patients who require full-dose anticoagulation (according to local guidelines). No Vitamin K antagonist and other anticoagulation allowed; LMWH allowed only for prevention not for curative treatment.
* History of pneumonitis within the last 5 years
* Patients who are under judicial protection and patients who are legally institutionalized.
* Patients unable or unwilling to comply with protocol
* Previous enrolment in this trial (Part 1 or Part 2).
* Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, makes them an unreliable trial patient or unlikely to complete the trial.
* Women who are pregnant, nursing, or who plan to become pregnant in the trial

Part 2:

* Known hypersensitivity to the trial drugs or their excipients or risk of allergic of anaphylactic reaction to drug product according to Investigator judgement (e.g. patient with history of anaphylactic reaction or autoimmune disease that is not controlled by nonsteroidal anti-inflammatory drugs (NSAIDs), inhaled corticosteroids, or the equivalent of </= 10 mg/day prednisone).
* Not more than one CPI based treatment regimen prior to entering study (e.g. anti-Programmed Death receptor-1 (PD-1), anti-Programmed Death-1 ligand-1 (PD-L1), anti-PD-L2, or anti-cytotoxic T lymphocyte associated antigen-4 (anti-CTLA-4) antibody). In case of CPIs combination, they need to be approved by the local regulatory agencies; for e.g., Melanoma cohort (Cohort E).
* Known HIV infection
* Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection (exception for patients in HCC cohorts; Cohorts F& G).
* History of severe hypersensitivity reactions to other mAbs.
* Immunosuppressive corticosteroid doses (> 10 mg prednisone daily or equivalent) within 4 weeks prior to the first dose of trial medication except for control of cerebral edema in case of recurrent glioblastoma (cohort D).
* Current or prior treatment with any systemic anti-cancer therapy (including radiotherapy) either within 28 days or a minimum of 5 half-lives, whichever is shorter before start of treatment
* Serious concomitant disease, especially those affecting compliance with trial requirements or which are considered relevant for the evaluation of the endpoints of the trial drug, such as neurologic, psychiatric, infectious disease or active ulcers (gastrointestinal tract, skin) or laboratory abnormality that may increase the risk associated with trial participation or trial drug administration, and in the judgment of the investigator would make the patient inappropriate for entry into the trial.
* Major injuries and/or surgery or bone fracture within 4 weeks of start of treatment, or planned surgical procedures during the trial period.
* Patients with personal or family history of QT prolongation and/or long QT syndrome, or prolonged QTcF at baseline (> 480 ms).
* Significant cardiovascular/cerebrovascular diseases (i.e. uncontrolled hypertension, unstable angina, history of infarction within past 6 months, congestive heart failure > NYHA II).

Uncontrolled hypertension defined as: Blood pressure in rested and relaxed condition >= 140 mmHg, systolic or >= 90 mmHg diastolic (with or without medication), measured according to Appendix 10.2.

* LVEF < 50%
* History of severe hemorrhagic or thromboembolic event in the past 12 months (excluding central venous catheter thrombosis and peripheral deep vein thrombosis).
* Known inherited predisposition to bleeding or to thrombosis in the opinion of the investigator.
* Patient with brain metastases that are symptomatic and/or require therapy.
* Patients who require full-dose anticoagulation (according to local guidelines).
* No Vitamin K antagonist and other anticoagulation allowed; LMWH allowed only for prevention not for curative treatment.
* History of pneumonitis (non-infectious) within the last 5 years
* Patients who are under judicial protection and patients who are legally institutionalized.
* Patients unable or unwilling to comply with protocol
* Previous enrolment in this trial.
* Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, makes them an unreliable trial patient or unlikely to complete the trial.
* Women who are pregnant, nursing, or who plan to become pregnant in the trial
* UncontrolledSymptomatic pleural effusion, pericardial effusion, or ascites
* Prior treatment with any antiangiogenic treatment (e.g. bevacizumab, cediranib, aflibercept, vandetanib, XL-184, sunitinib, etc) except for sorafenib and lenvatinib in 2nd line HCC cohort (Cohort F)
* Has received a live vaccine within 30 days prior to the first dose of study drug
* Patients with known active second malignancy other than non-melanoma skin cancers, non-metastatic prostate cancer, in situ cervical cancer, and ductal or lobular carcinoma in situ of the breast. Patients are not considered to have a currently active malignancy if they have completed anticancer therapy and have been disease free for greater than 2 years prior to screening
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-09-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (43):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Winship Cancer Institute, Atlanta, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
- Australia (4):
  - Royal North Shore Hospital-St Leonards-20807, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Peninsula & South Eastern Oncology Group, Frankston, Victoria
  - Alfred Hospital, Melbourne, Victoria
- France (6):
  - CTR Georges-François Leclerc, Dijon
  - HOP Timone, Marseille
  - INS Curie, Paris
  - CTR Eugène Marquis, Rennes
  - HOP Nord Laennec, Saint-Herblain
  - HOP Civil, Strasbourg
- Germany (5):
  - Universitätsklinikum Augsburg, Augsburg
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Regensburg, Regensburg
- Queen Mary Hospital, Hong Kong, Hong Kong
- Poland (5):
  - University Clinical Center, Gdansk, Gdansk
  - Mandziuk Slawomir Specialist Medical Practice, Lublin
  - European Health Center Otwock, Otwock
  - MED POLONIA SP Z O O, Clinical Trials Department,Poznan, Poznan
  - Dom Lekarski S.A., Szczecin
- Russia (3):
  - JSC "Group of Companies "Medsi", Moscow
  - SBHI "Saint-Petersburg Clinical Research Center of Specialized Types of Medical Care (Oncological)", Saint Petersburg
  - State Budget Healthcare Institution "Volgograd Regional Clinical Oncology Dispensary", Volgograd
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (3):
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Clinico Universitario De Valencia, Valencia
- Taiwan (2):
  - NCKUH, Tainan
  - National Taiwan University Hospital, Taipei
- Ukraine (4):
  - Municipal Non-profit Enterprise "City Clinical Hospital #4" of Dnipro City Council, Dnipropetrovks
  - Kyiv City Clinical Oncological Center, Kyiv
  - Medical and Preventive Treatment Inst. Volyn Regional, Lutsk, Lutsk
  - Vinnytsia Regional Clinical Oncological Dispensary, Vinnytsia
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-randomised, uncontrolled, open-label, dose escalating trial of BI 836880 administered in combination with ezabenlimab intravenously every 3 weeks. The trial consisted of 2 parts: Part 1 (dose escalation of BI 836880 in combination with ezabenlimab) and Part 2 (expansion phase in 8 cohorts).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Part 1 - BI 836880 360 mg | Part 1 - BI 836880 500 mg | Part 1 - BI 836880 720 mg | Part 2 - Cohort A, 2nd line NSCLC | Part 2 - Cohort B, 3rd line NSCLC | Part 2 - Cohort C, SCLC | Part 2 - Cohort D, glioblastoma | Part 2 - Cohort E, Melanoma | Part 2 - Cohort F, 2nd line Hepatocellular Carcinoma | Part 2 - Cohort G, 1st line Hepatocellular Carcinoma (HCC) | Part 2 - Cohort H, 2nd line HCC - atezolizumab in combination with bevacizumab failures
Started | 3 | 3 | 8 | 42 | 40 | 31 | 31 | 32 | 30 | 31 | 1
Completed (Subjects will on treatment.) | 0 | 1 | 0 | 6 | 5 | 3 | 2 | 1 | 6 | 2 | 0
Not Completed | 3 | 2 | 8 | 36 | 35 | 28 | 29 | 31 | 24 | 29 | 1
Not completed — Progressive disease | 3 | 0 | 4 | 20 | 23 | 15 | 24 | 27 | 13 | 13 | 0
Not completed — Other adverse event or clinical progression | 0 | 1 | 3 | 14 | 10 | 8 | 5 | 4 | 6 | 11 | 0
Not completed — Refused to continue taking trial medication | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 1 | 0 | 0
Not completed — Other than listed | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 4 | 4 | 1
Not completed — Dose Limiting Toxicity (DLT) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — missing reason | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This patient set includes all patients enrolled in the trial who were documented to have received at least one dose of ezabenlimab or BI 836880.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 - BI 836880 360 mg | Part 1 - BI 836880 500 mg | Part 1 - BI 836880 720 mg | Part 2 - Cohort A, 2nd Line NSCLC | Part 2 - Cohort B, 3rd Line NSCLC | Part 2 - Cohort C, SCLC | Part 2 - Cohort D, Glioblastoma | Part 2 - Cohort E, Melanoma | Part 2 - Cohort F, 2nd Line Hepatocellular Carcinoma | Part 2 - Cohort G, 1st Line Hepatocellular Carcinoma (HCC) | Part 2 - Cohort H, 2nd Line HCC - Atezolizumab in Combination With Bevacizumab Failures | Total
Number analyzed (Participants) | 3 | 3 | 8 | 42 | 40 | 31 | 31 | 32 | 30 | 31 | 1 | 252
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.3 (9.5) | 60.3 (2.1) | 58.3 (12.1) | 64.3 (9.1) | 59.2 (10.1) | 63.1 (11.7) | 56.7 (9.5) | 59.9 (14.7) | 64.4 (8.8) | 63.6 (9.4) | 55 (na) — not calculable with one subject | 61.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 15 | 18 | 10 | 10 | 10 | 4 | 7 | 1 | 80
  Male | 2 | 2 | 5 | 27 | 22 | 21 | 21 | 22 | 26 | 24 | 0 | 172
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 1 | 2 | 5 | 29 | 17 | 25 | 26 | 15 | 20 | 31 | 1 | 172
  Unknown or Not Reported | 2 | 1 | 3 | 13 | 23 | 5 | 4 | 16 | 10 | 0 | 0 | 77
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 10 | 3 | 4 | 6 | 4 | 8 | 4 | 0 | 39
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 2 | 5 | 19 | 14 | 24 | 20 | 12 | 12 | 25 | 1 | 135
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3 | 13 | 23 | 3 | 4 | 16 | 10 | 0 | 0 | 75

OUTCOME MEASURES:

1. Secondary Outcome: Part 1 - Adverse Events (AEs)
Description: The number of patients with any adverse events (AEs).
Time Frame: Up to 1263 days.
Population: All patients enrolled in part 1 of the trial who were documented to have received at least one dose of ezabenlimab or BI 836880.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1 - total: All patients in part 1 Patients received BI 836880 and 240 mg Ezabenlimab (BI 754091) as an intravenous infusion on day 1 of each 3-week cycle until progression, unacceptable toxicity, or up to a maximum of 53 cycles.
Arm/Group | Part 1 - BI 836880 360 mg | Part 1 - BI 836880 500 mg | Part 1 - BI 836880 720 mg | Part 1 - total
Number analyzed (Participants) | 3 | 3 | 8 | 14
Participants | 3 | 3 | 8 | 14

2. Secondary Outcome: Part 1 - Drug Related AEs
Description: The number of patients with any drug related adverse events (AEs).
Time Frame: Up to 1263 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 - BI 836880 360 mg | Part 1 - BI 836880 500 mg | Part 1 - BI 836880 720 mg | Part 1 - total
Number analyzed (Participants) | 3 | 3 | 8 | 14
Participants | 3 | 2 | 7 | 12

3. Secondary Outcome: Part 1 - Drug Related AEs Leading to Dose Reduction or Discontinuation
Description: The number of patients with any drug related adverse events (AEs) leading to dose reduction or discontinuation.
Time Frame: Up to 1263 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 - BI 836880 360 mg | Part 1 - BI 836880 500 mg | Part 1 - BI 836880 720 mg | Part 1 - total
Number analyzed (Participants) | 3 | 3 | 8 | 14
Participants
  Subjects with AEs leading to dose reduction of trial drug | 0 | 0 | 0 | 0
  Subjects with AEs leading to discontinuation of trial drug | 1 | 1 | 2 | 4

4. Secondary Outcome: Part 2 - Adverse Events (AEs)
Description: The number of patients with any adverse events (AEs).
Time Frame: Up to 778 days.
Population: All patients enrolled in part 2 of the trial who were documented to have received at least one dose of ezabenlimab or BI 836880.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2 - Cohort G, 1st line Hepatocellular Carcinoma: Patient with locally advanced or metastatic and/or unresectable HCC with no prior systemic treatment. This will be implemented only in countries where this cohort is approved. Patients received 720 milligram (mg) BI 836880 and 240 mg Ezabenlimab (BI 754091) as an intravenous infusion on day 1 of each 3-week cycle until progression, unacceptable toxicity, or up to a maximum of 53 cycles.
- Part 2 - total: All patients in part 2. Patients received 720 milligram (mg) BI 836880 and 240 mg Ezabenlimab (BI 754091) as an intravenous infusion on day 1 of each 3-week cycle until progression, unacceptable toxicity, or up to a maximum of 53 cycles.
Arm/Group | Part 2 - Cohort A, 2nd line NSCLC | Part 2 - Cohort B, 3rd line NSCLC | Part 2 - Cohort C, SCLC | Part 2 - Cohort D, glioblastoma | Part 2 - Cohort E, Melanoma | Part 2 - Cohort F, 2nd line Hepatocellular Carcinoma | Part 2 - Cohort G, 1st line Hepatocellular Carcinoma | Part 2 - Cohort H, 2nd line HCC - atezolizumab in combination with bevacizumab failures | Part 2 - total
Number analyzed (Participants) | 42 | 40 | 31 | 31 | 32 | 30 | 31 | 1 | 238
Participants | 39 | 39 | 27 | 30 | 31 | 28 | 28 | 1 | 223

5. Secondary Outcome: Part 2 - Drug Related AEs
Description: The number of patients with any drug related adverse events (AEs).
Time Frame: Up to 778 days.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 - Cohort A, 2nd line NSCLC | Part 2 - Cohort B, 3rd line NSCLC | Part 2 - Cohort C, SCLC | Part 2 - Cohort D, glioblastoma | Part 2 - Cohort E, Melanoma | Part 2 - Cohort F, 2nd line Hepatocellular Carcinoma | Part 2 - Cohort G, 1st line Hepatocellular Carcinoma | Part 2 - Cohort H, 2nd line HCC - atezolizumab in combination with bevacizumab failures | Part 2 - total
Number analyzed (Participants) | 42 | 40 | 31 | 31 | 32 | 30 | 31 | 1 | 238
Participants | 27 | 27 | 16 | 24 | 18 | 27 | 20 | 1 | 160

6. Secondary Outcome: Part 2 - Drug Related AEs Leading to Dose Reduction or Discontinuation
Description: The number of patients with any drug related adverse events (AEs) leading to dose reduction or discontinuation.
Time Frame: Up to 778 days.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 - Cohort A, 2nd line NSCLC | Part 2 - Cohort B, 3rd line NSCLC | Part 2 - Cohort C, SCLC | Part 2 - Cohort D, glioblastoma | Part 2 - Cohort E, Melanoma | Part 2 - Cohort F, 2nd line Hepatocellular Carcinoma | Part 2 - Cohort G, 1st line Hepatocellular Carcinoma | Part 2 - Cohort H, 2nd line HCC - atezolizumab in combination with bevacizumab failures | Part 2 - total
Number analyzed (Participants) | 42 | 40 | 31 | 31 | 32 | 30 | 31 | 1 | 238
Participants
  Subjects with AEs leading to dose reduction of trial drug | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3
  Subjects with AEs leading to discontinuation of trial drug | 13 | 4 | 6 | 2 | 2 | 5 | 6 | 0 | 38

7. Secondary Outcome: Part 2 - Disease Control (DC)
Description: Disease control (DC), defined as best overall response of CR, PR, or stable disease (SD) (Response Assessment in Neuro-Oncology (RANO for GBM & RECIST1.1 for all other cohorts).
Time Frame: Up to 778 days.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 - Cohort A, 2nd line NSCLC | Part 2 - Cohort B, 3rd line NSCLC | Part 2 - Cohort C, SCLC | Part 2 - Cohort D, glioblastoma | Part 2 - Cohort E, Melanoma | Part 2 - Cohort F, 2nd line Hepatocellular Carcinoma | Part 2 - Cohort G, 1st line Hepatocellular Carcinoma | Part 2 - Cohort H, 2nd line HCC - atezolizumab in combination with bevacizumab failures | Part 2 - total
Number analyzed (Participants) | 42 | 40 | 31 | 31 | 32 | 30 | 31 | 1 | 238
Participants | 34 | 25 | 12 | 25 | 18 | 24 | 25 | 1 | 164

8. Secondary Outcome: Part 2 - Duration of Objective Response (DoR)
Description: Duration of objective response (DoR), defined as the time from first documented CR or PR (RANO for GBM & RECIST1.1 for all other cohorts) until the earliest of disease progression or death among patients with OR.
Time Frame: Up to 84.4 weeks.
Population: All patients with an objective response enrolled in part 2 of the trial who were documented to have received at least one dose of ezabenlimab or BI 836880.
Measure: Median (Full Range); unit: weeks
Arm/Group | Part 2 - Cohort A, 2nd line NSCLC | Part 2 - Cohort B, 3rd line NSCLC | Part 2 - Cohort C, SCLC | Part 2 - Cohort D, glioblastoma | Part 2 - Cohort E, Melanoma | Part 2 - Cohort F, 2nd line Hepatocellular Carcinoma | Part 2 - Cohort G, 1st line Hepatocellular Carcinoma | Part 2 - Cohort H, 2nd line HCC - atezolizumab in combination with bevacizumab failures | Part 2 - total
Number analyzed (Participants) | 7 | 3 | 6 | 7 | 2 | 12 | 8 | 0 | 45
weeks | 23.4 [7.6 to 65.3] | 54.0 [48.4 to 58.0] | 30.0 [12.0 to 73.1] | 18.1 [10.7 to 78.3] | 43.3 [19.3 to 67.3] | 53.8 [6.3 to 84.4] | 48.9 [12.3 to 78.1] |  | 48.3 [6.3 to 84.4]

9. Secondary Outcome: Part 2 - Progression-free Survival (PFS)
Description: Progression-free survival (PFS) (RANO for GBM & RECIST1.1 for all other cohorts), defined as the time from first treatment infusion until disease progression or death from any cause, whichever occurs earlier. Tumour shrinkage (in millimeters), defined as the difference between the minimum post-baseline sum of diameters of target lesions (longest for non-nodal lesions, short axis for nodal lesions) and the baseline sum of diameters of the same set of target lesions in case of RECIST. In GBM, using RANO criteria, tumor shrinkage will be calculated based on the difference between the post-baseline and baseline measurements of the sum of product of the largest bi-dimensional measurements for all target lesions.
Time Frame: Up to 778 days.
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Part 2 - Cohort A, 2nd line NSCLC | Part 2 - Cohort B, 3rd line NSCLC | Part 2 - Cohort C, SCLC | Part 2 - Cohort D, glioblastoma | Part 2 - Cohort E, Melanoma | Part 2 - Cohort F, 2nd line Hepatocellular Carcinoma | Part 2 - Cohort G, 1st line Hepatocellular Carcinoma | Part 2 - Cohort H, 2nd line HCC - atezolizumab in combination with bevacizumab failures | Part 2 - total
Number analyzed (Participants) | 42 | 40 | 31 | 31 | 32 | 30 | 31 | 1 | 238
weeks | 43.14 [15.14 to 72.29] | 20.43 [7.29 to NA] — Not enough events reached to calculate the upper limit. | 6.29 [5.29 to 44.71] | 16.43 [11.43 to 59.86] | 27.86 [6.64 to 47.71] | 78.14 [11.86 to NA] — Not enough events reached to calculate the upper limit. | 37.00 [9.14 to 67.14] | 17.86 [17.86 to 17.86] | 28.00 [8.86 to 72.00]

10. Secondary Outcome: Part 1 - Maximum Measured Concentration of BI 836880 in Plasma (Cmax) After the First Infusion Cycle
Description: Part 1 - Maximum measured concentration of BI 836880 in plasma (Cmax) after the first infusion cycle.
Time Frame: 5 minutes before infusion and 1, 2.25, 6, 24, 168, 336 and 504 hours following the end of infusion in the first cycle.
Population: PK analysis set (PKS) part 1: This patient set included all patients in part 1 of the trial in the treated set who provide at least one evaluable observation for at least one PK endpoint and no PK relevant protocol deviation. Only subjects with available data were included, subjects were excluded due to various reasons, e.g., sample time deviations, deviations in dose or dosing time or too high predose concentrations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter
Arm/Group | Part 1 - BI 836880 360 mg | Part 1 - BI 836880 500 mg | Part 1 - BI 836880 720 mg
Number analyzed (Participants) | 0 | 1 | 3
microgram/milliliter |  | NA (na) — not disclosed due to data protection. | 175 (21.4)

11. Secondary Outcome: Part 1 - Maximum Measured Concentration of BI 836880 in Plasma (Cmax) After the Fourth Infusion Cycle
Description: Part 1 - Maximum measured concentration of BI 836880 in plasma (Cmax) after the fourth infusion cycle.
Time Frame: 5 minutes before infusion and 1, 2.25, 6, 24, 168, 336 and 504 hours following the end of infusion in the fourth cycle.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter
Arm/Group | Part 1 - BI 836880 360 mg | Part 1 - BI 836880 500 mg | Part 1 - BI 836880 720 mg
Number analyzed (Participants) | 0 | 1 | 4
microgram/milliliter |  | NA (na) — not disclosed due to data protection. | 273 (20.9)

12. Secondary Outcome: Part 1 - Time From Dosing to Maximum Serum Concentration of BI 836880 (Tmax) After the First Infusion Cycle
Description: Part 1 - Time from dosing to maximum serum concentration of BI 836880 (Tmax) after the first infusion cycle.
Time Frame: 5 minutes before infusion and 1, 2.25, 6, 24, 168, 336 and 504 hours following the end of infusion in the first cycle.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 1 - BI 836880 360 mg | Part 1 - BI 836880 500 mg | Part 1 - BI 836880 720 mg
Number analyzed (Participants) | 0 | 1 | 3
hours |  | NA (na) — not disclosed due to data protection. | 1.84 (134)

13. Secondary Outcome: Part 1 - Time From Dosing to Maximum Serum Concentration of BI 836880 (Tmax) After the Fourth Infusion Cycle
Description: Part 1 - Time from dosing to maximum serum concentration of BI 836880 (Tmax) after the fourth infusion cycle.
Time Frame: 5 minutes before infusion and 1, 2.25, 6, 24, 168, 336 and 504 hours following the end of infusion in the fourth cycle.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 1 - BI 836880 360 mg | Part 1 - BI 836880 500 mg | Part 1 - BI 836880 720 mg
Number analyzed (Participants) | 0 | 1 | 4
hours |  | NA (na) — not disclosed due to data protection. | 3.29 (91.9)

14. Secondary Outcome: Part 1 - Area Under the Concentration-time Curve of BI 836880 in Plasma Over the Time Interval From 0 to 504 Hours (AUC0-504h) After the First Infusion Cycle
Description: Part 1 - Area under the concentration-time curve of BI 836880 in plasma over the time interval from 0 to 504 hours (AUC0-504h) after the first infusion cycle.
Time Frame: 5 minutes before infusion and 1, 2.25, 6, 24, 168, 336 and 504 hours following the end of infusion in the first cycle.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*microgram/milliliter
Arm/Group | Part 1 - BI 836880 360 mg | Part 1 - BI 836880 500 mg | Part 1 - BI 836880 720 mg
Number analyzed (Participants) | 0 | 2 | 4
hours*microgram/milliliter |  | 19200 (28.5) | 35100 (20.9)

15. Secondary Outcome: Part 1 - Area Under the Concentration-time Curve of BI 836880 in Plasma Over the Time Interval From 0 to 504 Hours (AUC0-504h) After the Fourth Infusion Cycle
Description: Part 1 - Area under the concentration-time curve of BI 836880 in plasma over the time interval from 0 to 504 hours (AUC0-504h) after the fourth infusion cycle.
Time Frame: 5 minutes before infusion and 1, 2.25, 6, 24, 168, 336 and 504 hours following the end of infusion in the fourth cycle.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*microgram/milliliter
Arm/Group | Part 1 - BI 836880 360 mg | Part 1 - BI 836880 500 mg | Part 1 - BI 836880 720 mg
Number analyzed (Participants) | 0 | 1 | 4
hours*microgram/milliliter |  | NA (na) — not disclosed due to data protection. | 59700 (14.2)

16. Secondary Outcome: Part 2 - Maximum Measured Concentration of BI 836880 in Plasma (Cmax) After the First Infusion Cycle
Description: Part 2 - Maximum measured concentration of BI 836880 in plasma (Cmax) after the first infusion cycle.
Time Frame: 5 minutes before infusion and 1, 2.25, 6, 24, 168, 336 and 504 hours following the end of infusion in the first cycle.
Population: PK analysis set (PKS) part 2: This patient set included all patients in part 2 of the trial in the treated set who provide at least one evaluable observation for at least one PK endpoint and no PK relevant protocol deviation. Only subjects with available data were included, subjects were excluded due to various reasons, e.g., sample time deviations, deviations in dose or dosing time or too high predose concentrations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter
Arm/Group | Part 2 - Cohort A, 2nd line NSCLC | Part 2 - Cohort B, 3rd line NSCLC | Part 2 - Cohort C, SCLC | Part 2 - Cohort D, glioblastoma | Part 2 - Cohort E, Melanoma | Part 2 - Cohort F, 2nd line Hepatocellular Carcinoma | Part 2 - Cohort G, 1st line Hepatocellular Carcinoma | Part 2 - Cohort H, 2nd line HCC - atezolizumab in combination with bevacizumab failures
Number analyzed (Participants) | 38 | 38 | 29 | 30 | 25 | 30 | 25 | 1
microgram/milliliter | 251 (25.5) | 239 (30.5) | 275 (39.8) | 253 (23.4) | 240 (27.2) | 214 (20.5) | 206 (31.7) | NA (na) — not disclosed due to data protection.

17. Secondary Outcome: Part 2 - Time From Dosing to Maximum Serum Concentration of BI 836880 (Tmax) After the First Infusion Cycle
Description: Part 2 - Time from dosing to maximum serum concentration of BI 836880 (Tmax) after the first infusion cycle.
Time Frame: 5 minutes before infusion and 1, 2.25, 6, 24, 168, 336 and 504 hours following the end of infusion in the first cycle.
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 2 - Cohort A, 2nd line NSCLC | Part 2 - Cohort B, 3rd line NSCLC | Part 2 - Cohort C, SCLC | Part 2 - Cohort D, glioblastoma | Part 2 - Cohort E, Melanoma | Part 2 - Cohort F, 2nd line Hepatocellular Carcinoma | Part 2 - Cohort G, 1st line Hepatocellular Carcinoma | Part 2 - Cohort H, 2nd line HCC - atezolizumab in combination with bevacizumab failures
Number analyzed (Participants) | 38 | 38 | 29 | 30 | 25 | 30 | 25 | 1
hours | 2.75 (72.0) | 2.61 (91.6) | 2.25 (76.9) | 2.18 (73.9) | 2.47 (76.7) | 3.08 (109) | 2.54 (113) | NA (na) — not disclosed due to data protection.

18. Secondary Outcome: Part 2 - Area Under the Concentration-time Curve of BI 836880 in Plasma Over the Time Interval From 0 to 504 Hours (AUC0-504h) After the First Infusion Cycle
Description: Part 2 - Area under the concentration-time curve of BI 836880 in plasma over the time interval from 0 to 504 hours (AUC0-504h) after the first infusion cycle.
Time Frame: 5 minutes before infusion and 1, 2.25, 6, 24, 168, 336 and 504 hours following the end of infusion in the first cycle.
Population: PK analysis set (PKS) part 2: This patient set included all patients in part 2 of the trial in the treated set who provide at least one evaluable observation for at least one PK endpoint and no PK relevant protocol deviation, subjects were excluded due to various reasons, e.g., sample time deviations, deviations in dose or dosing time or too high predose concentrations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*microgram/milliliter
Arm/Group | Part 2 - Cohort A, 2nd line NSCLC | Part 2 - Cohort B, 3rd line NSCLC | Part 2 - Cohort C, SCLC | Part 2 - Cohort D, glioblastoma | Part 2 - Cohort E, Melanoma | Part 2 - Cohort F, 2nd line Hepatocellular Carcinoma | Part 2 - Cohort G, 1st line Hepatocellular Carcinoma | Part 2 - Cohort H, 2nd line HCC - atezolizumab in combination with bevacizumab failures
Number analyzed (Participants) | 35 | 32 | 18 | 28 | 28 | 24 | 24 | 1
hours*microgram/milliliter | 44000 (28.2) | 41300 (31.1) | 42000 (11.1) | 44900 (22.4) | 38000 (23.8) | 39400 (21.4) | 36600 (25.2) | NA (na) — not disclosed due to data protection.

19. Secondary Outcome: Part 1 - Maximum Measured Concentration of Ezabenlimab in Plasma (Cmax) After the First Infusion Cycle
Description: Part 1 - Maximum measured concentration of ezabenlimab in plasma (Cmax) after the first infusion cycle.
Time Frame: 5 minutes before infusion and 1, 2.25, 6, 24, 168, 336 and 504 hours following the end of infusion in the first cycle.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter
Arm/Group | Part 1 - BI 836880 360 mg | Part 1 - BI 836880 500 mg | Part 1 - BI 836880 720 mg
Number analyzed (Participants) | 3 | 2 | 7
microgram/milliliter | 80.7 (24.8) | 144 (78.9) | 75.8 (25.3)

20. Secondary Outcome: Part 1 - Maximum Measured Concentration of Ezabenlimab in Plasma (Cmax) After the Fourth Infusion Cycle
Description: Part 1 - Maximum measured concentration of ezabenlimab in plasma (Cmax) after the fourth infusion cycle.
Time Frame: 5 minutes before infusion and 1, 2.25, 6, 24, 168, 336 and 504 hours following the end of infusion in the fourth cycle.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter
Arm/Group | Part 1 - BI 836880 360 mg | Part 1 - BI 836880 500 mg | Part 1 - BI 836880 720 mg
Number analyzed (Participants) | 1 | 2 | 6
microgram/milliliter | NA (na) — not disclosed due to data protection. | 131 (16.2) | 106 (20.4)

21. Secondary Outcome: Part 1 - Time From Dosing to Maximum Serum Concentration of Ezabenlimab (Tmax) After the First Infusion Cycle
Description: Part 1 - Time from dosing to maximum serum concentration of ezabenlimab (Tmax) after the first infusion cycle.
Time Frame: 5 minutes before infusion and 1, 2.25, 6, 24, 168, 336 and 504 hours following the end of infusion in the first cycle.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 1 - BI 836880 360 mg | Part 1 - BI 836880 500 mg | Part 1 - BI 836880 720 mg
Number analyzed (Participants) | 3 | 2 | 7
hours | 1.83 (137) | 1.06 (7.84) | 2.79 (101)

22. Secondary Outcome: Part 1 - Time From Dosing to Maximum Serum Concentration of Ezabenlimab (Tmax) After the Fourth Infusion Cycle
Description: Part 1 - Time from dosing to maximum serum concentration of ezabenlimab (Tmax) after the fourth infusion cycle.
Time Frame: 5 minutes before infusion and 1, 2.25, 6, 24, 168, 336 and 504 hours following the end of infusion in the fourth cycle.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 1 - BI 836880 360 mg | Part 1 - BI 836880 500 mg | Part 1 - BI 836880 720 mg
Number analyzed (Participants) | 1 | 2 | 6
hours | NA (na) — not disclosed due to data protection. | 1.55 (65.5) | 2.32 (55.6)

23. Secondary Outcome: Part 1 - Area Under the Concentration-time Curve of Ezabenlimab in Plasma Over the Time Interval From 0 to 504 Hours (AUC0-504h) After the First Infusion Cycle
Description: Part 1 - Area under the concentration-time curve of ezabenlimab in plasma over the time interval from 0 to 504 hours (AUC0-504h) after the first infusion cycle.
Time Frame: 5 minutes before infusion and 1, 2.25, 6, 24, 168, 336 and 504 hours following the end of infusion in the first cycle.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*microgram/milliliter
Arm/Group | Part 1 - BI 836880 360 mg | Part 1 - BI 836880 500 mg | Part 1 - BI 836880 720 mg
Number analyzed (Participants) | 3 | 2 | 7
hours*microgram/milliliter | 15100 (42.0) | 15800 (8.13) | 14900 (27.5)

24. Secondary Outcome: Part 1 - Area Under the Concentration-time Curve of Ezabenlimab in Plasma Over the Time Interval From 0 to 504 Hours (AUC0-504h) After the Fourth Infusion Cycle
Description: Part 1 - Area under the concentration-time curve of ezabenlimab in plasma over the time interval from 0 to 504 hours (AUC0-504h) after the fourth infusion cycle.
Time Frame: 5 minutes before infusion and 1, 2.25, 6, 24, 168, 336 and 504 hours following the end of infusion in the fourth cycle.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*microgram/milliliter
Arm/Group | Part 1 - BI 836880 360 mg | Part 1 - BI 836880 500 mg | Part 1 - BI 836880 720 mg
Number analyzed (Participants) | 1 | 2 | 5
hours*microgram/milliliter | NA (na) — not disclosed due to data protection. | 34000 (17.8) | 25200 (32.5)

25. Secondary Outcome: Part 2 - Maximum Measured Concentration of Ezabenlimab in Plasma (Cmax) After the First Infusion Cycle
Description: Part 2 - Maximum measured concentration of ezabenlimab in plasma (Cmax) after the first infusion cycle.
Time Frame: 5 minutes before infusion and 1, 2.25, 6, 24, 168, 336 and 504 hours following the end of infusion in the first cycle.
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter
Arm/Group | Part 2 - Cohort A, 2nd line NSCLC | Part 2 - Cohort B, 3rd line NSCLC | Part 2 - Cohort C, SCLC | Part 2 - Cohort D, glioblastoma | Part 2 - Cohort E, Melanoma | Part 2 - Cohort F, 2nd line Hepatocellular Carcinoma | Part 2 - Cohort G, 1st line Hepatocellular Carcinoma | Part 2 - Cohort H, 2nd line HCC - atezolizumab in combination with bevacizumab failures
Number analyzed (Participants) | 41 | 38 | 28 | 29 | 27 | 28 | 29 | 1
microgram/milliliter | 85.7 (26.3) | 80.5 (22.0) | 89.3 (27.8) | 87.7 (22.3) | 76.6 (18.2) | 74.6 (20.1) | 71.3 (28.3) | NA (na) — not disclosed due to data protection.

26. Secondary Outcome: Part 2 - Time From Dosing to Maximum Serum Concentration of Ezabenlimab (Tmax) After the First Infusion Cycle
Description: Part 2 - Time from dosing to maximum serum concentration of ezabenlimab (Tmax) after the first infusion cycle.
Time Frame: 5 minutes before infusion and 1, 2.25, 6, 24, 168, 336 and 504 hours following the end of infusion in the first cycle.
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 2 - Cohort A, 2nd line NSCLC | Part 2 - Cohort B, 3rd line NSCLC | Part 2 - Cohort C, SCLC | Part 2 - Cohort D, glioblastoma | Part 2 - Cohort E, Melanoma | Part 2 - Cohort F, 2nd line Hepatocellular Carcinoma | Part 2 - Cohort G, 1st line Hepatocellular Carcinoma | Part 2 - Cohort H, 2nd line HCC - atezolizumab in combination with bevacizumab failures
Number analyzed (Participants) | 41 | 38 | 28 | 29 | 27 | 28 | 29 | 1
hours | 2.93 (129) | 2.90 (68.2) | 2.26 (77.8) | 2.35 (84.8) | 3.03 (65.9) | 2.38 (63.8) | 2.75 (110) | NA (na) — not disclosed due to data protection.

27. Secondary Outcome: Part 2 - Area Under the Concentration-time Curve of Ezabenlimab in Plasma Over the Time Interval From 0 to 504 Hours (AUC0-504h) After the First Infusion Cycle
Description: Part 2 - Area under the concentration-time curve of ezabenlimab in plasma over the time interval from 0 to 504 hours (AUC0-504h) after the first infusion cycle.
Time Frame: 5 minutes before infusion and 1, 2.25, 6, 24, 168, 336 and 504 hours following the end of infusion in the first cycle.
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*microgram/milliliter
Arm/Group | Part 2 - Cohort A, 2nd line NSCLC | Part 2 - Cohort B, 3rd line NSCLC | Part 2 - Cohort C, SCLC | Part 2 - Cohort D, glioblastoma | Part 2 - Cohort E, Melanoma | Part 2 - Cohort F, 2nd line Hepatocellular Carcinoma | Part 2 - Cohort G, 1st line Hepatocellular Carcinoma | Part 2 - Cohort H, 2nd line HCC - atezolizumab in combination with bevacizumab failures
Number analyzed (Participants) | 36 | 34 | 17 | 30 | 31 | 25 | 26 | 1
hours*microgram/milliliter | 17600 (29.7) | 15200 (35.2) | 17700 (16.9) | 19300 (22.1) | 14500 (25.5) | 14900 (23.1) | 14200 (31.5) | NA (na) — not disclosed due to data protection.

28. Primary Outcome: Part 1 - Number of Patients With Dose Limiting Toxicity (DLT) Within the First Cycle of Treatment
Description: Number of patients with dose limiting toxicity (DLT) within the first cycle of treatment.
Time Frame: The first treatment cycle, up to 21 days.
Population: Maximum tolerated dose (MTD) set: This patient set includes all patients enrolled in dose escalation and confirmation of MTD cohort of the trial (Part 1) who were documented to have received at least one dose of ezabenlimab or BI 836880 and were evaluable for the MTD determination.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 - BI 836880 360 mg | Part 1 - BI 836880 500 mg | Part 1 - BI 836880 720 mg | Part 1 - total
Number analyzed (Participants) | 3 | 3 | 8 | 14
Participants | 1 | 0 | 0 | 1

29. Primary Outcome: Part 2 - Objective Response (OR)
Description: Objective Response (OR) defined as best overall response (Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1)) of complete response (CR) or partial response (PR) from first treatment infusion until the earliest of disease progression, death or last evaluable tumor assessment before start of subsequent anticancer therapy, lost to follow-up, or withdrawal of consent. In case of recurrent glioblastoma (GBM), assessment will be based on RANO (Response Assessment in Neuro-Oncology) criteria.
Time Frame: Up to 778 days.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 - Cohort A, 2nd line NSCLC | Part 2 - Cohort B, 3rd line NSCLC | Part 2 - Cohort C, SCLC | Part 2 - Cohort D, glioblastoma | Part 2 - Cohort E, Melanoma | Part 2 - Cohort F, 2nd line Hepatocellular Carcinoma | Part 2 - Cohort G, 1st line Hepatocellular Carcinoma | Part 2 - Cohort H, 2nd line HCC - atezolizumab in combination with bevacizumab failures | Part 2 - total
Number analyzed (Participants) | 42 | 40 | 31 | 31 | 32 | 30 | 31 | 1 | 238
Participants | 7 | 3 | 6 | 7 | 2 | 12 | 8 | 0 | 45

ADVERSE EVENTS:
Time Frame: From the start of treatment until the end of treatment + 42 days of residual effect period, up to 1263 days.
Description: Treated set (TS): This patient set includes all patients enrolled in the trial who were documented to have received at least one dose of ezabenlimab or BI 836880.
Arm/Group | Part 1 - BI 836880 360 mg | Part 1 - BI 836880 500 mg | Part 1 - BI 836880 720 mg | Part 2 - Cohort A, 2nd line NSCLC | Part 2 - Cohort B, 3rd line NSCLC | Part 2 - Cohort C, SCLC | Part 2 - Cohort D, glioblastoma | Part 2 - Cohort E, Melanoma | Part 2 - Cohort F, 2nd line Hepatocellular Carcinoma | Part 2 - Cohort G, 1st line Hepatocellular Carcinoma | Part 2 - Cohort H, 2nd line HCC - atezolizumab in combination with bevacizumab failures
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/3 | 1/8 | 4/42 | 2/40 | 5/31 | 1/31 | 2/32 | 4/30 | 5/31 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 6/8 | 24/42 | 21/40 | 14/31 | 10/31 | 11/32 | 16/30 | 17/31 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 8/8 | 36/42 | 35/40 | 23/31 | 28/31 | 30/32 | 28/30 | 27/31 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 - BI 836880 360 mg (N=3) | Part 1 - BI 836880 500 mg (N=3) | Part 1 - BI 836880 720 mg (N=8) | Part 2 - Cohort A, 2nd line NSCLC (N=42) | Part 2 - Cohort B, 3rd line NSCLC (N=40) | Part 2 - Cohort C, SCLC (N=31) | Part 2 - Cohort D, glioblastoma (N=31) | Part 2 - Cohort E, Melanoma (N=32) | Part 2 - Cohort F, 2nd line Hepatocellular Carcinoma (N=30) | Part 2 - Cohort G, 1st line Hepatocellular Carcinoma (N=31) | Part 2 - Cohort H, 2nd line HCC - atezolizumab in combination with bevacizumab failures (N=1)
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 1 | 0
Stoma site cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 1 | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device breakage (Product issues) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Hyperthermia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ill-defined disorder (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Perforated ulcer (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spontaneous bacterial peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coma scale abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paraneoplastic myelopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Thrombosis in device (Product issues) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Autoimmune nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelocaliectasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 2 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Embolism venous (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral venous disease (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 - BI 836880 360 mg (N=3) | Part 1 - BI 836880 500 mg (N=3) | Part 1 - BI 836880 720 mg (N=8) | Part 2 - Cohort A, 2nd line NSCLC (N=42) | Part 2 - Cohort B, 3rd line NSCLC (N=40) | Part 2 - Cohort C, SCLC (N=31) | Part 2 - Cohort D, glioblastoma (N=31) | Part 2 - Cohort E, Melanoma (N=32) | Part 2 - Cohort F, 2nd line Hepatocellular Carcinoma (N=30) | Part 2 - Cohort G, 1st line Hepatocellular Carcinoma (N=31) | Part 2 - Cohort H, 2nd line HCC - atezolizumab in combination with bevacizumab failures (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 5 | 5 | 0 | 0 | 3 | 2 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 4 | 1 | 2 | 4 | 2 | 5 | 6 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 5 | 1 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 2 | 6 | 5 | 4 | 1 | 4 | 4 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 3 | 11 | 4 | 4 | 3 | 9 | 9 | 5 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 3 | 12 | 14 | 8 | 9 | 10 | 7 | 3 | 0
Chest pain (General disorders) | 0 | 2 | 0 | 3 | 4 | 2 | 0 | 1 | 2 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 3 | 3 | 6 | 4 | 4 | 3 | 4 | 5 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 5 | 4 | 2 | 4 | 3 | 9 | 4 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 3 | 1 | 2 | 1 | 0 | 1 | 3 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 2 | 3 | 3 | 4 | 1 | 4 | 5 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 4 | 8 | 3 | 3 | 2 | 5 | 4 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 4 | 6 | 0 | 2 | 2 | 3 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 1 | 5 | 9 | 0 | 2 | 1 | 2 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 9 | 8 | 4 | 0 | 9 | 5 | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3 | 4 | 2 | 0 | 2 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 3 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 5 | 2 | 3 | 3 | 5 | 8 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 3 | 3 | 1 | 4 | 3 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2 | 3 | 0 | 1 | 0 | 3 | 2 | 0
Headache (Nervous system disorders) | 0 | 2 | 1 | 4 | 4 | 1 | 4 | 4 | 5 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1 | 7 | 2 | 5 | 3 | 2 | 13 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 9 | 7 | 5 | 0 | 4 | 6 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 6 | 8 | 7 | 0 | 4 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 5 | 2 | 3 | 2 | 3 | 7 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 5 | 1 | 1 | 4 | 2 | 2 | 0
Hypertension (Vascular disorders) | 2 | 2 | 5 | 10 | 9 | 4 | 8 | 4 | 13 | 4 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Hyperleukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 3 | 3 | 1 | 0 | 4 | 1 | 0 | 0
Monocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Neutrophilia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 0 | 3 | 6 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 3 | 0 | 0
Eye discharge (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 5 | 2 | 0 | 1 | 3 | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 3 | 8 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 4 | 6 | 8 | 4 | 4 | 5 | 2 | 2 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 4 | 6 | 3 | 3 | 1 | 3 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Hyperthermia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 3 | 1 | 1 | 4 | 3 | 1 | 3 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 4 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 2 | 0 | 3 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 5 | 4 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth avulsion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 1 | 3 | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 0 | 2 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 2 | 8 | 3 | 1 | 1 | 0 | 2 | 4 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 1 | 0 | 10 | 0 | 1 | 1 | 1 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 3 | 5 | 0 | 3 | 3 | 1 | 2 | 0
Blood triglycerides increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 4 | 4 | 0 | 0 | 4 | 1 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 4 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Platelet count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Weight decreased (Investigations) | 0 | 1 | 1 | 2 | 1 | 3 | 1 | 1 | 1 | 3 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 4 | 1 | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 5 | 4 | 0 | 0 | 0 | 0 | 2 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 4 | 8 | 0 | 1 | 2 | 3 | 3 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 2 | 2 | 0 | 2 | 0 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 5 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 1 | 1 | 1 | 2 | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 2 | 2 | 2 | 1 | 1 | 1 | 1 | 0
Monoparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 1 | 3 | 1 | 0 | 1 | 1 | 2 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Distractibility (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 2 | 3 | 3 | 2 | 3 | 1 | 2 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ketonuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 4 | 3 | 0 | 2 | 2 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 2 | 1 | 0 | 2 | 1 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
White coat hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-05-18): https://cdn.clinicaltrials.gov/large-docs/26/NCT03468426/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/26/NCT03468426/SAP_001.pdf